CLINICAL TRIAL: NCT03476798
Title: A Phase II Trial of Bevacizumab and Rucaparib in Recurrent Carcinoma of the Cervix or Endometrium
Brief Title: Bevacizumab and Rucaparib in Recurrent Carcinoma of the Cervix or Endometrium
Acronym: Clovis-001
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Oklahoma (Other)
Collaborators: Clovis Oncology, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: OU-SCC-CLOVIS-001
Record Dates: First submitted 2018-03-19; First posted 2018-03-26 (Actual); Results first posted 2021-05-28 (Actual); Last update posted 2024-02-15 (Actual); Status verified 2024-02

CONDITIONS: Cervical Cancer; Endometrial Cancer
MeSH Terms: conditions — Uterine Cervical Neoplasms; Endometrial Neoplasms | interventions — rucaparib; Bevacizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Bevacizumab + Rucaparib (Experimental)
  Interventions: Drug: Rucaparib; Drug: Bevacizumab

INTERVENTIONS:
Drug: Rucaparib — Rucaparib 600mg PO BID daily
Drug: Bevacizumab — Bevacizumab 15mg/kg IV on day 1 of each cycle

SUMMARY:
This is a phase II study of rucaparib, a small molecule inhibitor poly (adenosine diphosphate [ADP]-ribose) polymerase (PARP), being tested in combination with bevacizumab in patients with recurrent cervical or endometrial cancer. The objective of this study is to determine the proportion of these patients who survive progression-free for at least 6 months while receiving this drug combination.

DETAILED DESCRIPTION:
Patients who consent to participate in this study will receive treatment with rucaparib and bevacizumab until unacceptable toxicity or tumor progression. Subjects will take one rucaparib pill will be taken twice daily, and bevacizumab will be adimistered via IV onDay 1 of each 21 day cycle. Subjects will receive tests and procedures that are part of regular cancer care as well as those required for the purposes of this study. If there is no cancer found in scans after 6 cycles of treatment, patients may continue with study treatment for 1 year. Follow up visits will occur every 3 months for the first 2 years after treatment is completed and every 6 months for 3 additional years.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with histologically-documented carcinoma of the cervix or endometrium.
2. Patients with measurable and/or evaluable lesions as defined by RECIST 1.1.
3. Women at least 18 years of age
4. Patients with persistent or recurrent squamous cell or adenocarcinoma of the cervix, or any carcinoma or carcinosarcoma of the endometrium who has undergone at least one prior line of systemic therapy. Prior bevacizumab is allowed. (Note: previous cisplatin during radiation therapy should NOT count as a prior line of systemic therapy).
5. ECOG performance status of 0, 1, or 2.
6. Patients should agree to have tumor biopsy for correlative studies.If the patients are unable to be safely biopsied and desire enrollment, they may be enrolled per principal investigator discretion.
7. Adequate organ function should be confirmed by the following laboratory values obtained ≤ 14 days prior to first dose of rucaparib.
8. Patients must have a life expectancy of at least 3 months ((to be able to complete one cycle of study treatment).
9. Patients should have no major existing co-morbidities or medical conditions that will preclude therapy in the view of the principal investigator.
10. Prior bevacizumab is allowed if off drug ≥ 28 days prior to study enrollment.
11. Women of childbearing potential must not be considering getting pregnant and must avoid pregnancy during the study and for at least six months after the last dose of rucaparib or longer if requested by local authorities.

Exclusion Criteria:

1. Have active second malignancy, i.e., patient known to have potentially fatal cancer present for which she may be (but not necessarily) currently receiving treatment; However patients with a history of malignancy that has been completely treated, with no evidence of that cancer currently, are permitted to enroll in the trial provided all chemotherapy was completed >6 months prior and/or bone marrow transplant (BMT) >2 years prior to first dose of rucaparib.
2. Prior treatment with any PARP inhibitor.
3. Untreated or symptomatic central nervous system (CNS) metastases.Patients with asymptomatic CNS metastases are eligible provided they have been clinically stable for at least 4 weeks.
4. Patients who have received treatment with chemotherapy within 4 weeks (6 weeks for nitrosoureas or mitomycin C); or radiation, biologic/targeted agents, experimental drugs within 3 weeks prior to first dose of rucaparib; and/or ongoing adverse effects from such treatment > NCI CTCAE Grade 1 (Grade 2 non-hematologic toxicity to most recent treatment may be permitted with prior advanced approval from Sponsor).
5. Hospitalization for bowel obstruction within 3 months prior to enrollment.
6. Patients must have no history of gross hemoptysis (defined as bright red blood of a ½ teaspoon or more) or coagulopathy. Patients with history of major tumor-related bleeding that is not controlled despite locoregional treatment or at high risk of recurrent tumor-related bleeding will be excluded.
7. Patients with history of hypertension must be well-controlled (≤150/100) on a stable regimen of anti-hypertensive therapy.
8. Patients with tumors that invaded major vessels (e.g. the carotid) as shown unequivocally by imaging studies will be excluded due to the possibility of increased risk for tumor bleeding with bevacizumab therapy.
9. Patients should not have a major surgical procedure, open biopsy, or significant traumatic injury within 28 days prior to study enrollment, or anticipation of need for major surgical procedure during the course of the study. No history of abdominal fistula, gastrointestinal perforation, or intra-abdominal abscess within 28 days prior to registration. No serious non-healing wound, ulcer, or bone fracture.
10. Patients should not have unstable angina or myocardial infarction within the previous 6 months; no uncontrolled hypertension; no symptomatic congestive heart failure; no serious cardiac arrhythmia requiring medication; no clinically significant peripheral vascular disease; no history of any CNS cerebrovascular ischemia or stroke within the last 6 months; no active serious infection.
11. Patients should not have other coexisting medical condition that would preclude full compliance with the study.
12. Patients may not be receiving any other investigational agents.
13. Patients should not have a history of prior severe infusion reaction to a monoclonal antibody. Patients with known hypersensitivity of Chinese hamster ovary cell products or other recombinant human antibodies.
14. Pregnant women are excluded from this study because rucaparib and bevacizumab have the potential for teratogenic or abortifacient effects. Because there is an unknown but potential risk for adverse events in nursing infants secondary to treatment of the mother with rucaparib and bevacizumab, breastfeeding should be discontinued if the mother is treated with rucaparib and bevacizumab. Should a woman become pregnant or suspect she is pregnant while in this study, she should inform her treating physician immediately.
15. HIV-positive patients receiving combination anti-retroviral therapy are excluded from the study because of possible drug interactions with rucaparib and bevacizumab.

Ages: 18 Years to 99 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 49 (Actual)
Dates: Start 2018-06-29 (Actual); Primary Completion 2020-05-12 (Actual); Study Completion 2023-09-29 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kathleen Moore, MD, Principal Investigator — Obstetrics and Gynecology
Locations (3):
- United States (3):
  - University of Minnesota, Minneapolis, Minnesota
  - Stephenson Cancer Center, University of Oklahoma Health Sciences Center, Oklahoma City, Oklahoma
  - University of Virginia Cancer Center, Charlottesville, Virginia

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited at 3 cancer centers from June 2018 to Nov 2019. The first patient was enrolled on July 2, 2018 and the last patient was enrolled on November 8, 2019
Pre-assignment Details: Of 49 enrolled participants, 33 met inclusion criteria and assign to the single arm treatment. Among 33 participants started treatment, 28 were evaluable for statistical analysis.
Period: Overall Study
Arm/Group | Bevacizumab + Rucaparib
Started | 33
Completed | 28
Not Completed | 5
Not completed — Death | 1
Not completed — Withdrawal by Subject | 2
Not completed — Protocol Violation | 2

BASELINE CHARACTERISTICS:
Arm/Group | Bevacizumab + Rucaparib
Number analyzed (Participants) | 33
Age, Continuous [Mean (Standard Deviation); unit: years] | 60.4 (12.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 33
  Male | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1
  Not Hispanic or Latino | 32
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 2
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 4
  White | 27
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 33

OUTCOME MEASURES:

1. Primary Outcome: Proportion of Patients Who Are Progression-free at 6 Months
Description: To estimate the proportion of pts treated w/bevacizumab who are progression-free.
  Progression for measurable disease per RECIST v1.1. Progression for pts with non-measurable disease at baseline is defined as increasing clinical, radiological, or histological evidence of disease since study entry.
Time Frame: 6 months
Population: Patients who met criteria for evaluability: Evaluable patients will be defined as patients with measurable and/or evaluable lesions who received at least cycle 1 doses of study treatment (one dose of IV bevacizumab and 21 days of rucaprib, PO, BID) and complete the first post-treatment CT or MRI for tumor assessment.
Measure: Number (95% Confidence Interval); unit: Proportion of patients
Arm/Group | Bevacizumab + Rucaparib
Number analyzed (Participants) | 28
Proportion of patients | 0.29 [0.13 to 0.47]

2. Secondary Outcome: Proportion of Patients Who Had Objective Tumor Response
Description: To estimate the proportion of patients treated with bevacizumab and rucaparib who have objective tumor response (complete or partial)
Time Frame: up to 2 years
Measure: Number (95% Confidence Interval); unit: Proportion of patients
Arm/Group | Bevacizumab + Rucaparib
Number analyzed (Participants) | 28
Proportion of patients | 0.14 [0.04 to 0.33]

3. Secondary Outcome: Number of Patients Who Experience Toxicity
Description: To determine the nature and degree of toxicity in combination of rucaparib and bevacizumab (Adverse Event Grade 3 and higher).
Time Frame: up to 2 year
Population: All patients who received treatment
Measure: Count of Participants; unit: Participants
Arm/Group | Bevacizumab + Rucaparib
Number analyzed (Participants) | 33
Participants | 22

4. Secondary Outcome: Median Overall Survival
Description: To estimate the median overall survival of patients treated with combination rucaparib and bevacizumab.
Time Frame: up to 2 years
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Bevacizumab + Rucaparib
Number analyzed (Participants) | 28
Months | 10.12 [7.04 to 15.17]

5. Secondary Outcome: Median Progression-free Survival Time
Description: To estimate the progression-free survival (PFS) of patients with persistent or recurrent cervical or endometrial cancer treated with combination rucaparib and bevacizumab Progression for measurable disease per RECIST v1.1 Progression for patients with non-measurable disease at baseline is defined as increasing clinical, radiological, or histological evidence of disease since study entry.
Time Frame: up to 2 years
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Bevacizumab + Rucaparib
Number analyzed (Participants) | 28
Months | 3.83 [2.51 to 5.72]

ADVERSE EVENTS:
Time Frame: up to 34 months
Arm/Group | Bevacizumab + Rucaparib
All-Cause Mortality (participants affected / at risk) | 29/33
Serious Adverse Events (participants affected / at risk) | 14/33
Other Adverse Events (participants affected / at risk) | 33/33
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Bevacizumab + Rucaparib (N=33)
Abdominal pain (Gastrointestinal disorders) | 2
Nausea (Gastrointestinal disorders) | 4
Vomiting (Gastrointestinal disorders) | 4
Fatigue (General disorders) | 2
Sepsis (Infections and infestations) | 2
Urinary tract infection (Infections and infestations) | 2
Acute kidney injury (Renal and urinary disorders) | 3
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 2
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 2
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Bevacizumab + Rucaparib (N=33)
Anemia (Blood and lymphatic system disorders) | 8
Sinus tachycardia (Cardiac disorders) | 2
Blurred vision (Eye disorders) | 3
Abdominal pain (Gastrointestinal disorders) | 4
Constipation (Gastrointestinal disorders) | 8
Diarrhea (Gastrointestinal disorders) | 16
Gastroesophageal reflux disease (Gastrointestinal disorders) | 4
Mucositis oral (Gastrointestinal disorders) | 6
Nausea (Gastrointestinal disorders) | 21
Vomiting (Gastrointestinal disorders) | 16
Edema limbs (General disorders) | 2
Fatigue (General disorders) | 19
Fever (General disorders) | 4
Localized edema (General disorders) | 8
Pain (General disorders) | 5
Otitis externa (Infections and infestations) | 2
Sinusitis (Infections and infestations) | 3
Urinary tract infection (Infections and infestations) | 9
Bruising (Injury, poisoning and procedural complications) | 5
Alanine aminotransferase increased (Investigations) | 5
Alkaline phosphatase increased (Investigations) | 3
Aspartate aminotransferase increased (Investigations) | 5
Blood bilirubin increased (Investigations) | 5
Blood lactate dehydrogenase increased (Investigations) | 2
Cholesterol high (Investigations) | 3
Creatinine increased (Investigations) | 6
Platelet count decreased (Investigations) | 7
Weight loss (Investigations) | 7
Anorexia (Metabolism and nutrition disorders) | 9
Hyperglycemia (Metabolism and nutrition disorders) | 2
Hyperkalemia (Metabolism and nutrition disorders) | 2
Hypoalbuminemia (Metabolism and nutrition disorders) | 3
Hypocalcemia (Metabolism and nutrition disorders) | 2
Hypokalemia (Metabolism and nutrition disorders) | 3
Hypomagnesemia (Metabolism and nutrition disorders) | 2
Hyponatremia (Metabolism and nutrition disorders) | 2
Arthralgia (Musculoskeletal and connective tissue disorders) | 6
Back pain (Musculoskeletal and connective tissue disorders) | 4
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 2
Myalgia (Musculoskeletal and connective tissue disorders) | 8
Dizziness (Nervous system disorders) | 11
Dysgeusia (Nervous system disorders) | 8
Headache (Nervous system disorders) | 15
Peripheral sensory neuropathy (Nervous system disorders) | 3
Agitation (Psychiatric disorders) | 7
Anxiety (Psychiatric disorders) | 4
Hematuria (Renal and urinary disorders) | 4
Proteinuria (Renal and urinary disorders) | 10
Urinary frequency (Renal and urinary disorders) | 4
Vaginal hemorrhage (Reproductive system and breast disorders) | 3
Cough (Respiratory, thoracic and mediastinal disorders) | 11
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 8
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 7
Alopecia (Skin and subcutaneous tissue disorders) | 3
Dry skin (Skin and subcutaneous tissue disorders) | 9
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 5
Hot flashes (Vascular disorders) | 5
Hypertension (Vascular disorders) | 19
Hypotension (Vascular disorders) | 2
Thromboembolic event (Vascular disorders) | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (3):
  • Study Protocol (2020-04-01): https://cdn.clinicaltrials.gov/large-docs/98/NCT03476798/Prot_000.pdf
  • Statistical Analysis Plan (2021-05-03): https://cdn.clinicaltrials.gov/large-docs/98/NCT03476798/SAP_001.pdf
  • Informed Consent Form (2020-02-19): https://cdn.clinicaltrials.gov/large-docs/98/NCT03476798/ICF_002.pdf